CLINICAL TRIAL: NCT03961152
Title: Effect of the PainCoach App on Pain and Opiate Use in the First Two Weeks After Total Knee Replacement: Randomised Controlled Trial
Brief Title: Effect of the PainCoach App on Pain and Opiate Use After Total Knee Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kliniek ViaSana (Other)
Collaborators: St. Anna Ziekenhuis, Geldrop, Netherlands (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: PainCoach app study
Record Dates: First submitted 2019-05-14; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Total Knee Replacement; Pain; Opioid Use; E-health App
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: Patients were randomised to the PainCoach-app group or control group. Both groups received usual care. In the PainCoach-app group, in addition to receiving the aforementioned usual care, patients could use the PainCoach app whenever they wanted. In response to the patient's input of the pain experienced, the app gave advice on pain medication use, exercises/rest and when to call the clinic. This advice was the same as patients also received during usual care.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PainCoach-app group (Experimental): In the PainCoach-app group, in addition to receiving the aforementioned usual care, the PainCoach app was downloaded on each patient's smartphone or tablet. Patients could use this app whenever they wanted until day 14 after surgery. They were not subjected to any different treatment compared to the control group, i.e. advice on pain management was delivered in an extra and different way, but the pain medication itself was exactly the same for both groups.
  Interventions: Behavioral: PainCoach app
- Control group (No Intervention): The control group received usual care.

INTERVENTIONS:
Behavioral: PainCoach app — In response to the patient's input of the pain experienced (no pain, bearable pain, unbearable pain, or untenable pain), the app gave advice on pain medication use, exercises/rest and when to call the clinic from day 1 until day 14 after surgery.
  Arms: PainCoach-app group

SUMMARY:
Less is known about pain and opiate use at home directly after total knee replacement (TKR). Regarding side effects, low opiate use is desired. An e-health application, PainCoach app, was developed to guide patients in pain control and opiate use.

The aim of this study was to investigate the effect of the PainCoach app on pain and opiate use in TKR patients in the first two weeks at home after surgery. The hypothesis was that the use of this app would decrease pain and opiate use.

ELIGIBILITY:
Inclusion Criteria:

* Planned for primary TKR

Exclusion Criteria:

* No possession of a smartphone or tablet
* Contra-indication to any of the pain medication used in the study
* No email address
* No internet at home
* No thorough command of the Dutch language
* Suffering from memory disorders
* Surgery under general anaesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2017-06-08 (Actual)

PRIMARY OUTCOMES:
Change in pain at rest in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  Pain at rest was daily measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Change in pain during activity in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  Measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Change in pain at night in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  Measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Change in opiate use in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  Oxycodon (5 mg per tablet) use was recorded in quantities per 24 hours

SECONDARY OUTCOMES:
Pain at rest | 1 month after surgery
  Measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Pain during activity | 1 month after surgery
  Measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Pain at night | 1 month after surgery
  Measured with VAS from 0 (no pain) to 100 (worst imaginable pain)
Change in other pain medication use in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  i.e. NSAID (Diclofenac), acetaminophen and/or Gabapentin were recorded in quantities per 24 hours
Change in pain acceptance at rest, during activity and at night in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14, and at 1 month after surgery
  Measured with a happy smiley (acceptable pain) and a sad smiley (unacceptable pain)
Change in experiences with the executed recommended physiotherapy exercises in the first two weeks at home after TKR | 14 measurement points: daily from day 1 to 14 after surgery
  Measured on a 3-item scale; did too much, exactly enough, or could have done more exercises
Function | 1 month after surgery
  Measured with the Knee injury and Osteoarthritis Outcome Score - Physical Function Short-form (KOOS-PS) with a total score from 0 (no difficulty) to 100 (extreme difficulty)
Function and pain | 1 month after surgery
  Measured with the Oxford Knee Score (OKS) with a total score from 0 (most severe symptoms) to 48 (least severe symptoms)
Quality of life | 1 month after surgery
  Measured with the EuroQol-5D 3 level version (EQ-5D-3L) consisting of two scores: EQ Visual Analogue Scale (EQ VAS) score from 0 (worst imaginable health state) to 100 (best imaginable health state), and EQ-5D descriptive system (EQ-5D index).
PainCoach app's perceived effectiveness | Day 14 after surgery
  Usability, added value, and likelihood of being recommended to others was recorded on a 5-item scale ranging from totally agree to totally disagree
Active PainCoach app use | From day 1 to 14 after surgery
  Measured with recording the actual amount of app use and defining active use as at least 12 times in total

CONTACTS AND LOCATIONS:
Overall Officials: J.M. Brinkman, MD, PhD, Principal Investigator — Kliniek ViaSana
Locations (1):
- Kliniek ViaSana, Mill, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pronk Y, Peters MCWM, Sheombar A, Brinkman JM. Effectiveness of a Mobile eHealth App in Guiding Patients in Pain Control and Opiate Use After Total Knee Replacement: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2020 Mar 13;8(3):e16415. doi: 10.2196/16415. PMID 32167483